CLINICAL TRIAL: NCT03071822
Title: Combination Chemotherapy Including Cisplatin, Ifosfamide, Gemcitabine, L-asparaginase, Etoposide and Dexamethasone (PIGLETS Regimen) as Treatment of Newly Diagnosed and Relapsed/Refractory Peripheral T Cell Lymphomas (PTCLs)
Brief Title: Combination Chemotherapy Including Cisplatin, Ifosfamide, Gemcitabine, L-asparaginase, Etoposide and Dexamethasone as Treatment of Newly Diagnosed and Relapsed/Refractory Peripheral T Cell Lymphomas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yok-lam Kwong, Chair Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-001
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: PTCLs
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Cisplatin; Ifosfamide; Gemcitabine; Asparaginase; Etoposide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patient will be given this combination of chemotherapy (cisplatin, ifosfamide, gemcitabine, L-asparaginase, etoposide and dexamethasone) for a total of 6 courses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PIGLETs (Experimental): Patient will be given this combination of chemotherapy (cisplatin, ifosfamide, gemcitabine, L-asparaginase, etoposide and dexamethasone) for a total of 6 courses
  Interventions: Drug: cisplatin; Drug: ifosfamide; Drug: gemcitabine; Drug: L-asparaginase; Drug: etoposide; Drug: dexamethasone

INTERVENTIONS:
Drug: cisplatin — PIGLETs
Drug: ifosfamide — PIGLETs
Drug: gemcitabine — PIGLETs
Drug: L-asparaginase — PIGLETs
Drug: etoposide — PIGLETs
Drug: dexamethasone — PIGLETs

SUMMARY:
The PIGLETS regimen was devised to replace the conventional SMILE regimen in management of extranodal NK/T cell lymphoma in our institution. It had been three years since the introduction of PIGLETS regimen in treatment of NK malignancies. The response rate is encouraging, with an overall response rate (ORR) of 90% in NK malignancies. Side effects are generally tolerable. The investigator therefore propose the use of PIGLETS on newly diagnosed or relapsed/refractory PTCLs.

DETAILED DESCRIPTION:
Peripheral T cell lymphomas (PTCLs) are a group of heterogenous lymphoid malignancies derived from post-thymic mature T-lymphocytes. They are further classified according to their putative origin, immunophenotype, sites of involvement and clinical behaviour. Common subtypes include PTCL-not otherwise specified (PTCL-NOS), angioimmunoblastic T cell lymphoma (AITL) and anaplastic large cell lymphoma (ALCL). With the exception of ALCL, PTCLs behave aggressively and their response to chemotherapy is typically poor. CHOP regimen (cyclophosphamide, doxorubicin, vincristine, prednisolone) borrowed from treatment of B-cell lymphoma is commonly used. However, there is no randomized controlled trial evaluating its efficacy. Moreover, despite the initial response of 40-70%, most patients suffer from disease relapse, giving rise to disappointing five year disease free survival (DFS) and overall survival (OS), typically in the range of 30% and 20%, respectively. As a result, there is not yet a standard agreed-on regimen for treatment of PTCLs in an upfront setting.

One of the possible mechanisms behind the intrinsic resistance to chemotherapy in PTCLs is the overexpression of multi-drug resistance (MDR) gene/P-glycoprotein (P-gp), which mediates active efflux of chemotherapeutic medications out of intracellular compartment. Regimens combining drugs which are independent of the P-gp pathway were proven to be successful in the management of PTCL, extranodal NK/T cell lymphoma, a lymphoma also expressing high level of MDR gene/P-glycoprotein. The PIGLETS regimen was devised to replace the conventional SMILE regimen in management of extranodal NK/T cell lymphoma in our institution. It had been three years since the introduction of PIGLETS regimen in treatment of NK malignancies. The response rate is encouraging, with an overall response rate (ORR) of 90% in NK malignancies. Side effects are generally tolerable. The investigator therefore propose the use of PIGLETS on newly diagnosed or relapsed/refractory PTCLs.

Expected toxicity:

1. The PIGLETS regimen had been in used since 2013, with the toxicities well known to the investigators
2. Typical side effects of chemotherapy would be anticipated, including cytopenia, alopecia, mucositis and emesis. These can all be managed with supportive therapy
3. Anaphylactic reaction to L-asparaginase may occur, but a small test dose will be given before formal administration to ensure the absence of allergy. Prophylactic antihistamine and glucocorticoids will also be given.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age of 18 - 80 years, with confirmed PTCLs
2. Adequate organ functions
3. ECOG performance status of <=2
4. No history of hypersensitivity to any of the components of the PIGLETS regimen
5. Informed consent obtained

Exclusion Criteria:

1. Inadequate organ functions
2. ECOG performance status of >=3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events and severe adverse events | 1 year
  Incidence of AE and SAE by severity grading as assessed according to CTCAE v4.03
  Incidence of AE and SAE by severity grading as assessed according to CTCAE v4.03
Overall response rate (ORR) | 3 months
  proportion of patients achieving CR or CRi or partial remission (PR)
Overall response rate (ORR) | 6 months
  proportion of patients achieving CR or CRi or partial remission (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Yok Lam Kwong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong